CLINICAL TRIAL: NCT01983215
Title: EFFECTS OF PREVENA THERAPY ON REDUCTION OF GROIN SURGICAL SITE INFECTIONS IN OBESE PATIENTS UNDERGOING VASCULAR SURGERY
Brief Title: Effects of Prevena Therapy on Obese and or Diabetic Patients With Surgical Groin Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Jean E. Starr, MD (Other)
Responsible Party: Sponsor-Investigator, Dr. Jean E. Starr, MD, Vascular surgeon, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013H0045
Record Dates: First submitted 2013-09-27; First posted 2013-11-13 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Diabetes; Peripheral Vascular Disease
Keywords: groin incisions
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Peripheral Vascular Diseases | interventions — Random Allocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- negative pressure dressing vs. standard of care (Experimental): single arm study- randomized Prevena vac or standard of care
  Interventions: Device: Prevena vac

INTERVENTIONS:
Device: Prevena vac
  Other Names: randomized 1:1 negative pressure dressing vs. standard of care

SUMMARY:
The purpose of the study is to determine the effects of Prevena therapy on decreasing groin surgical site infections in patients who are obese and /or diabetic having vascular surgery.

DETAILED DESCRIPTION:
Patients who are obese and/or diabetic may have poor surgical healing and infection rates higher. The PREVENA therapy will be used to evaluate possible reduction of infection rates in this patient population

ELIGIBILITY:
Inclusion Criteria:

* subjects over 18 years old
* obese (BMI > 30) and or diabetic

Exclusion Criteria:

* current infected surgical field, hemodialysis, immunosuppressive therapy, allergy to adhesive, sensitivity to silver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2013-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with infections | 30 day post surgical procedure
  reduction of 30 day surgical site infection by evaluating infection rates in obese, diabetic patients who were randomized to Prevena Vac vs. standard of care

SECONDARY OUTCOMES:
infection rates | 1 year
  reduction of 1 year graft infection in prosthetic grafts and reduction of secondary hospitalizations for infection.Patients will be followed through 1 year to measure results of infection rates and secondary hospitalization related to infection

CONTACTS AND LOCATIONS:
Overall Officials: Jean E Starr, MD, Principal Investigator — The Ohio State Medical Center
Locations (1):
- Ohio State Division of Vascular Diseases and Surgery, Columbus, Ohio, United States